CLINICAL TRIAL: NCT01335113
Title: A Scan Ultrasonography in the Evaluation of Retinopathy of Prematurity
Status: Terminated | Type: Observational
Why Stopped: Unable to get accurate measurements with existing technology
Sponsor: Stanford University (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Darius M. Moshfeghi, Principle Investigator, Stanford University
Other Study IDs: 19891
Record Dates: First submitted 2011-04-01; First posted 2011-04-14 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the investigators study is to determine the relationship between the length of the eye and the rate of change in eye length at each visit with progression of retinopathy of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* neonates being screened for retinopathy of prematurity

Exclusion Criteria:

* medically unstable neonates

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature newborns who are screened for retinopathy of prematurity at Stanford
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
axial length | one year
  axial length as measured by a scan ulstrasonography

SECONDARY OUTCOMES:
anterior corneal curvature | one year
  anterior corneal curvature as measured by keratometer
wide angle fundus photography | one year
  wide angle fundus photography by RetCam camera

CONTACTS AND LOCATIONS:
Overall Officials: Darius M Moshfeghi, MD, Study Director — Stanford University; Darius Moshfeghi, MD, Principal Investigator — Stanford University
Locations (1):
- University of Miami, Miami, Florida, United States